CLINICAL TRIAL: NCT02198131
Title: Pulsed Dye Laser for Treatment of Post Radiation Dysphonia
Brief Title: Pulsed Dye Laser in Treating Patients With Post Radiation Dysphonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00011092; NCI-2014-01458 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98214 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Oral Complications of Radiation Therapy; Stage I Laryngeal Cancer; Stage II Laryngeal Cancer
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (pulsed dye laser) (Experimental): Patients undergo pulsed dye laser monthly for three months.
  Interventions: Procedure: laser therapy; Other: questionnaire administration

INTERVENTIONS:
Procedure: laser therapy — Undergo pulsed dye laser
  Other Names: therapy, laser
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot trial studies pulsed dye laser in treating patients with post radiation dysphonia. Dysphonia, or vocal cord scarring, can include trouble with the voice when trying to talk, such as hoarseness, change in voice pitch, and poor voice quality, and it commonly happens after radiation therapy for laryngeal cancer. Pulsed dye laser may improve post radiation dysphonia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the use of pulsed dye laser in treatment of the dysphonia that commonly results after radiation therapy for laryngeal carcinoma.

OUTLINE:

Patients undergo pulsed dye laser monthly for three months.

After completion of study treatment, patients are followed up at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from dysphonia after radiation therapy for glottic carcinoma will be included in the study
* Patients will be included if their initial stage was T1 N0 M0 or T2 N0 M0

Exclusion Criteria:

* Patients having previously undergone large surgical resections of the larynx or hypopharynx will be excluded
* Patients fewer than 1 year out from completion of radiation therapy will be excluded
* Patients with local disease recurrence would be excluded from the trial
* Patients in whom the transnasal endoscope is poorly tolerated or patients in whom transnasal endoscopic laryngoscopy is contraindicated will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Videostroboscopy rates | Up to 6 months post-treatment
  Forced choice comparisons will be utilized in the pre and post treatment stroboscopy comparisons.
Change in Voice Handicap Index (VHI)-10 score | Baseline to 6 months post-treatment
  The VHI-10 form will be scored and then those numbers will be compared pre and post treatment for each individual.
Change in jitter | Baseline and at 6 months post-treatment
  Laboratory based voice analysis will be performed with evaluations of aerodynamics and acoustics.
Voice quality using the patient self-assessment questionnaire | Up to 6 months post-treatment
  The post treatment questionnaire form will be scored and then comparisons made for each individual question on the form across our study group. These values will be discrete variables.
Change in shimmer | Baseline and at 6 months post-treatment
  Laboratory based voice analysis will be performed with evaluations of aerodynamics and acoustics.
Change in noise to harmonic ratio | Baseline and at 6 months post-treatment
  Laboratory based voice analysis will be performed with evaluations of aerodynamics and acoustics.
Change in mean phonatory flow | Baseline and at 6 months post-treatment
  Laboratory based voice analysis will be performed with evaluations of aerodynamics and acoustics.

CONTACTS AND LOCATIONS:
Overall Officials: Carter Wright, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States